CLINICAL TRIAL: NCT04593095
Title: Nurturing and Quiet Intervention (NeuroN-QI) on Preterm Infants' Neurodevelopment and Maternal Stress and Anxiety: Protocol of a Pilot Randomized Clinical Trial
Brief Title: Nurturing and Quiet Intervention: NeuroN-QI
Acronym: NeuroN-QI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Marilyn Aita, Associate Professor & Researcher, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MP-21-2020-2587 (MP)
Record Dates: First submitted 2020-08-25; First posted 2020-10-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-11

CONDITIONS: Neurodevelopment
Keywords: developmental care; preterm infants; mothers; pilot study

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Each SSC session will last 2-hr during the day including a 15-min of auditory stimulation with maternal voice and controlled levels of NICU light and noise. The 2-hr SSC will be followed by a 1-hr quiet period where infants will rest in their incubator/crib with a pad immersed with their mother breast milk for olfactory stimulation and where the control of light and noise levels will be continued. The NeuroN-QI will be done 4 times/wk for each dyad.
  Interventions: Other: NeuroN-QI
- Control (No Intervention): Mothers-infant dyads will do 4 SSC/wk. During these sessions, no attempt will be made by the RA to control the light and noise levels nor to encourage auditory stimulation. The SSC periods will not be followed by a quiet period nor olfactory stimulation.

INTERVENTIONS:
Other: NeuroN-QI — SSC session lasting 2-hr during the day 4 times/wk including a 15-min of auditory stimulation with maternal voice and controlled levels of NICU light and noise followed by a 1-hr quiet period where infants will rest in their incubator/crib with olfactory stimulation and where the control of light and noise levels will be continued.
  Arms: Experimental

SUMMARY:
The current state of knowledge reveals that the development of the brain of preterm infants is influenced by specific neonatal experiences during hospitalization, such as environmental sensory stimulation (light and noise), as well as physical and emotional proximity to mothers. However, there is a lack of evidence regarding the benefits that could be associated with the combination of care interventions to improve the health outcomes of preterm infants and their mothers, and in particular the development of the brain of infants during their hospitalization in the neonatal unit. The aim of this pilot study is to assess the feasibility and acceptability of a developmental care intervention including periods of nurturing between mothers and their infant (skin-to-skin contact and auditory stimulation) to promote physical and emotional proximity and a quiet period (controlled light and noise levels and olfactory stimulation in incubators) and to estimate the effect of this intervention on infants' neurodevelopment as well as on maternal stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

Infants:

- born between 26 and 316/7 WGA.

Mothers

* agree to do 4 SSC sessions/week with a 15-minutes period of auditory (reading) stimulation;
* express breast milk for their infant;
* speak, read, or write French or English.

Nurses:

* have at least 6 months of work experience in a NICU;
* speak and read French or English.

Exclusion Criteria:

Infants:

* have birth defects or genetic disorders;
* have an intraventricular hemorrhage > grade II;
* receive nasal respiratory support;
* have been transferred from another hospital.

Mothers:

* are <18 years of age;
* had a multiparous birth;
* have a physical condition that does not allow SSC;
* abuse substances or alcohol;
* do not intend to breastfeed or give breastmilk.

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the NeuroN-QI and the study procedures as assessed by a self-completed questionnaire (mothers) and a logbook (RA) | 1 year
  questionnaire completed by mothers - each question treated separately (no total score) Log book completed by a research assistant

SECONDARY OUTCOMES:
Estimated effects of NeuroN-QI on infants' neurodevelopment as assessed using the Assessment of Preterm Infants Behavior (APIB) | 1 year
  Observation scale by videos
Estimated effects of NeuroN-QI on infants' neurodevelopment as assessed using the General Movements Assessment (GMA) | 1 year
  Observation by videos
Estimated effects of NeuroN-QI on maternal stress as assessed by PSS:NICU | 1 year
Estimated effects of NeuroN-QI on maternal anxiety as assessed by STAI-Y | 1 year
Nurses' training needs about the NeuroN-QI as assessed by a self-completed questionnaire | 1 year
  Questionnaire completed by nurses - each question treated separately from strongly disagree to totally strongly agree (no total score)
Acceptability of the NeuroN-QI as assessed by a self-completed questionnaire | 1 year
  questionnaire completed by nurses - each question treated separately from totally acceptable to totally unacceptable (no total score)
Feasibility of the NeuroN-QI as assessed by a self-completed questionnaire | 1 year
  questionnaire completed by nurses - each question treated separately from totally feasible to totally unfeasible (no total score)

OTHER OUTCOMES:
Confounding variables | 1 year
  birth weight, WGA at birth, postnatal age at the beginning of the intervention, APGAR score, mothers' use of psychological health care resources, other SSC sessions, SNAPPE-II, and light and noise levels with soundmeter and light meter

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Aita, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aita M, Heon M, Lavallee A, De Clifford Faugere G, Altit G, Le May S, Dorval V, Lippe S, Larone Juneau A, Remmer E, Rennick JE. Nurturing and quiet intervention (NeuroN-QI) on preterm infants' neurodevelopment and maternal stress and anxiety: A pilot randomized clinical trial protocol. J Adv Nurs. 2021 Jul;77(7):3192-3203. doi: 10.1111/jan.14819. Epub 2021 Mar 14. PMID 33719093